CLINICAL TRIAL: NCT02467374
Title: Pilot: Fear Extinction and Mechanisms of Change in Obsessive Compulsive Disorder
Brief Title: Fear Extinction and Mechanisms of Change in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Sabine Wilhelm, PhD, Chief of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P002325
Record Dates: First submitted 2015-06-01; First posted 2015-06-10 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; Neuroimaging; Fear Extinction; Behavior Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Behavior Therapy (Active Comparator): If assigned to the immediate BT condition, patients will be asked to make about 24 visits to our clinics at MGH, including an initial assessment, 12 therapy visits over 12 weeks, and 1 booster session (Week 16). Patients will be asked to come to the clinic for assessments during weeks 4 and 6 and after the treatment (week 12), as well as 1 follow-up visit (week 24). Additionally, patients will participate in 6 MRI scanning sessions at the Charlestown Navy Yard.
  Interventions: Behavioral: Behavior Therapy
- Waitlist Behavior Therapy (Active Comparator): Patients will wait for 12 weeks before starting BT. In this case, they will be asked to make about 21 visits to our clinics, including an initial assessment visit, 12 therapy visits, and 1 booster session. Patients will be asked to come to the clinic for assessments during (weeks 4 and 6) and after the waiting period (week 12). Additionally, patients will participate in 6 MRI scanning sessions at the Charlestown Navy Yard.
  Interventions: Behavioral: Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy — BT for OCD focuses primarily on "exposure with response prevention (ERP)." "ERP" involves gradual exposure to anxiety-provoking situations (things or situations that frighten or disturb some people), and will help to prevent compulsions (repetitive behaviors).
  Other Names: Exposure and Response Prevention

SUMMARY:
The purpose of this study is to find out more about how the brain stores emotional learning in obsessive-compulsive disorder (OCD). In particular, we would like to understand how human beings learn not to fear. We are also interested in learning about how behavioral therapy (BT) for OCD affects emotional learning in the brain. We hope this study will help us understand why people with OCD cannot control unwanted fear and to develop better treatments for adults with OCD. Patients will be randomly assigned (like the flip of a coin) to receive 12 weeks of BT or 12 weeks of waitlist, followed by 12 weeks of BT. We are seeking individuals 18-60 with OCD and individuals with no psychiatric history. Participation includes a diagnostic evaluation, 12 weeks of BT or 12 weeks of waitlist followed by BT, questionnaires, and up to six (6) MRI scans. You may receive up to $500 for your participation and reimbursement for parking.

DETAILED DESCRIPTION:
The purpose of this study is to find out more about how the brain forms and stores emotional learning. Emotional learning refers to our ability to form an association between sounds or places with emotional events. In particular, we would like to understand how human beings learn not to fear and whether individuals with OCD use certain areas of the brain differently than control individuals. We hope this study will help us understand why people with OCD cannot control unwanted fear. We are also interested in learning about how behavioral therapy (BT) for OCD affects emotional learning in the brain. Patients in this study will have an equal chance of undergoing 12 weeks of BT immediately or being placed on a 12-week "waitlist," and then partaking in BT. They will be asked to participate in tasks while in an MRI that takes pictures of the brain. This study will also use mild, half-second electric shocks to fingers. The electric current will be generated from a 9V battery (e.g., battery in a smoke alarm). In order to set the level of the current to be used during the study, we will begin at a level below what patients will be able to feel, and then increase in gradual steps with permission. Patients will be asked to stop the increase at a level of the current that they find highly annoying but not painful. The level of current that patients select during this trial procedure, and no higher level, will be used during the study so that they will not receive any painful electric shocks. The purpose of the electric shock is to create a situation in which emotional learning may occur. Patients will receive no more than ten of these electric shocks.

If patients are assigned to immediate BT, participation in this study includes about 20-22 visits to our two clinics at MGH and the Charlestown Navy Yard over the span of 6 months. This includes an initial assessment visit (2.5-3 hours), 12 therapy visits (each session lasting 60-90 minutes long), and 1 booster session at the MGH OCD and Related Disorders Clinic. During the course of therapy, patients will receive weekly practice work between sessions, which should take around 30 minutes to an hour each day to complete. Additionally, patients will participate in 3 MRI scanning sessions at the Charlestown Navy Yard Campus: 2 scans over a two-day period during baseline visit, 2 scans over a two-day period during week 4 visit, and 2 scans over a two-day period during 3-month follow-up (week 24) appointment.

If patients are assigned to the 12-week waiting period before starting BT, participation will include about 21 visits to our clinics, including an initial assessment visit (2.5-3 hours), 12 therapy visits (after the waiting period ends), and 1 booster session at the MGH OCD and Related Disorders Clinic. Patients will be asked to come to the clinic for assessments during weeks 4 and 6 and after the waiting period (week 12). Patients will also participate in 2 MRI scanning sessions at the Charlestown Navy Yard Campus: 2 scans over a two-day period during baseline visit and 2 scans over a two-day period during week 4 visit. Patients may NOT begin any new therapy or medication while on the waiting list.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18 to 60, proficient in English, and able to give informed consent
* For OCD patients only: Primary OCD that causes at least moderate distress and/or impairment (Y-BOCS total score > 16)

Exclusion Criteria:

* Current clinically significant suicidality and/or BDI-II suicide item (#9) score >1
* Current or history of neurologic or psychiatric disease (e.g., mental retardation, dementia, brain damage, or other cognitive impairment) that would interfere with ability to engage in BT
* Psychopathology not appropriate for the treatment (such as substance abuse or dependence within the past 3 months; current manic episode; psychosis)
* Previous treatment with ≥4 sessions of BT for OCD
* Currently receiving any other psychotherapy or planning to initiate such treatment during the study
* Use of conventional antipsychotic medications or medications that would lower seizure threshold in high doses or may otherwise affect cerebral metabolism (other than to those required for stabilization of OCD).
* Use of benzodiazepines within 2 weeks prior to study is not allowed. Use of other psychotropic medications (e.g., SSRIs and atypical antipsychotics) will be allowed provided the dose has been stable for > 8 weeks. Planning on initiation or dose change of psychotropic medication during the study.
* Impaired (or uncorrected) vision, medical illness, or medical treatment that would likely interfere with participation.
* History of head injury resulting in prolonged loss of consciousness and/or neurological sequelae; History of seizures; History of stroke; Signs of increased intracranial pressure; Prior neurosurgical procedure
* Metal in the body, metal injury to the eyes; Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt
* Pregnancy; breastfeeding or nursing; if the patient cannot rule out the possibility of pregnancy, a pregnancy test (to be ruled out by urine ß-HCG) will be conducted prior to study
* Weight > 250 lbs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Obsessive compulsive symptoms as measured by Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 24-36 weeks
  We assesed reduction in OCD symptom severity over a 24 week period. Efficacy was again compared in the follow-up phase of the study in from week 24 to week 36.

OTHER OUTCOMES:
Fear Conditioning/Extinction Paradigm | 24-36 weeks
  Test Paradigm within MRI scanner
Skin Conductance | 24-36 weeks
  Recording electrodes will be attached to the palm of the subject's left hand to measure Skin Conductance Rate (SCR). SCR will be measured through a 9-mm (sensor diameter) Sensor Medics Ag/AgCl electrodes (safe for use in the magnet environment).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital: Department of Psychiatry; Mohammed Milad, Ph.D., Principal Investigator — Massachusetts General Hospital: Department of Psychiatry
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Jacoby RJ, Greenberg JL, Hurtado A, Pedersen W, Ellard KK, Pace-Schott EF, Oliver KI, Milad MR, Wilhelm S, Camprodon JA. Neural mechanisms underlying exposure and response prevention for obsessive compulsive disorder: A randomized controlled trial. Behav Res Ther. 2025 Nov;194:104858. doi: 10.1016/j.brat.2025.104858. Epub 2025 Sep 17. PMID 41005270